CLINICAL TRIAL: NCT04473079
Title: Efficacy and Safety of Lacidofil® STRONG as an Adjuvant for Helicobacter Pylori Eradication Treatment in Non-ulcer Dyspepsia: A Randomized, Placebo-controlled, Double-blind, Parallel Study
Brief Title: Efficacy and Safety of Lacidofil® STRONG as an Adjuvant for Helicobacter Pylori Treatment in Non-ulcer Dyspepsia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: I-020
Record Dates: First submitted 2020-07-09; First posted 2020-07-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-02

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): These participants will receive the standard treatment for H. pylori eradication (proton-pump inhibitor and antibiotics) plus probiotic formulation (commercially-available as Lacidofil) for 12 weeks.
  Interventions: Dietary Supplement: Lacidofil
- Placebo group (Placebo Comparator): These participants will receive the standard treatment for H. pylori eradication (proton-pump inhibitor and antibiotics) plus placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lacidofil — Investigational product intake daily for 6 weeks. Co-administration of H. pylori treatment with investigational product the first two weeks only.
  Arms: Experimental group
Dietary Supplement: Placebo — Investigational product intake daily for 6 weeks. Co-administration of H. pylori treatment with investigational product the first two weeks only.
  Arms: Placebo group

SUMMARY:
Treatment for H. pylori eradication includes antibiotics. The treatment has decreased its efficiency (lower capability to eradicate the infection) due to increasing antibiotic resistance in the population. But the addition of probiotics to the treatment has been observed to increase efficiency, and decreasing the antibiotics' side effects. We set to evaluate whether Lacidofil® STRONG improves efficacy when added to the standard therapy to eradicate H. pylori.

DETAILED DESCRIPTION:
This study aims at evaluating the efficacy of Lacidofil® STRONG as an adjuvant therapy to a standard 14-day H. pylori eradication treatment among H. pylori-positive participants with non-ulcer dyspepsia.

This is a randomized, placebo-controlled trial, with two parallel arms. Participants will be randomized to receive probiotic or placebo as adjuvant to the standard anti-H. pylori treatment. Each participant will be enrolled in the study for 12 weeks, during which they will receive the anti-H. pylori treatment and co-administration of investigational product (IP; for two weeks), followed by IP supplementation alone (for four weeks), and they will be followed-up 4 weeks after last IP administration.

ELIGIBILITY:
Inclusion Criteria:

* Thai patients consulting for dyspeptic symptoms.
* Aged between 18 and 65 years.
* Diagnosed for H. pylori infection using RUT and 13C-UBT.
* H. pylori treatment naïve.
* Able to provide informed consent.
* Willing to maintain their usual physical activity regime and diet, as well as discontinuing the consumption probiotic-containing and fermented foods.

Exclusion Criteria:

* Upper gastrointestinal bleeding.
* Presence of duodenal or gastric ulcers, MALT lymphoma, gastric resection, gastric malignancy as per endoscopy (visual assessment).
* Current intake of antibiotics, such as amoxicillin, clarithromycin, metronidazole or fluoroquinolone.
* Use of probiotics in the past month, and unwilling to undergo a 2-week washout period before the study.
* Use of NSAIDs, aspirin or other anti-inflammatory drugs within 1 week (for occasional use) or 3 weeks (for chronic use) of inclusion.
* Contraindication for gastric biopsy (e.g., coagulopathy).
* Any history of allergy for penicillin, levofloxacin, clarithromycin or rabeprazole.
* Receiving proton pump inhibitor within 4 weeks or receiving any antibiotics or bismuth within 2 weeks of trial initiation.
* Being pregnant or breastfeeding.
* Having severe underlying disease including end-stage renal disease requiring hemodialysis or peritoneal dialysis (GFR < 15), cirrhosis with Child-Pugh classification grade C, immuno-compromised host with AIDS, malignancy and/or cerebrovascular or cardiovascular disease.
* Taking anticoagulants (e.g., warfarin) or anti-platelet agents (e.g., clopidogrel)
* Previous gastric surgery.
* Having underlying heart disease, including congenital long QT syndrome.
* Unwilling to stop taking over-the-counter, natural or herbal medicines for dyspeptic or gastrointestinal symptoms (e.g., antidiarrheal, anti-emetics, antacids) during the intervention period (6 weeks).
* Milk and soy allergy.
* Lactose intolerance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Rate of H. pylori eradication | At week 6 after treatment
  Efficacy of the H. pylori eradication treatment supplemented with Lacidofil will be done by calculating the proportion of participants reaching H. pylori eradication in probiotics group compared to placebo, as per urea breath test (13C-UBT)
Rate of H. pylori eradication | At week 12 after treatment
  Efficacy of the H. pylori eradication treatment supplemented with Lacidofil will be done by calculating the proportion of participants reaching H. pylori eradication in probiotics group compared to placebo, as per urea breath test (13C-UBT)

SECONDARY OUTCOMES:
Efficacy: Frequency and severity of dyspeptic symptoms from baseline | At week 6 after treatment
  Evaluated by the administration of the Severity of Dyspepsia Assessment (SODA; ranges differ at all three scales) at the end of eradication treatment
Efficacy: Severity of gastrointestinal symptoms | At week 6 after treatment
  Evaluated by the administration of the Gastrointestinal Symptoms Rating Scale (GSRS; overall score range 0 - No discomfort to 105 - Very severe discomfort) at the end of eradication treatment
Efficacy: Health-related quality of life (HR-QoL) | At week 6 after treatment
  Evaluated by the administration of the 36-Item Short Form Survey Instrument (SF-36; score ranges 0 - worst possible health to 100 - best possible health) at the end of eradication treatment
Quantification of adverse events during the intervention | At week 12 after treatment
  Quantification of adverse and serious adverse events deemed by PI as related to the probiotic

CONTACTS AND LOCATIONS:
Overall Officials: Ratha-korn Vilaichone, Principal Investigator — Thammasat University Hospital
Locations (1):
- Thammasat University Hospital, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kiattiweerasak A, Aumpan N, Chonprasertsuk S, Pornthisarn B, Siramolpiwat S, Bhanthumkomol P, Nunanan P, Issariyakulkarn N, Mahachai V, Yamaoka Y and Vilaichone R-k. Efficacy and safety of Lacticaseibacillus rhamnosus R0011 and Lactobacillus helveticus R0052 as an adjuvant for Helicobacter pylori eradication: a double-blind, randomized, placebo-controlled study. Frontiers in Gastroenterology 2023; 2:1245993. doi: 10.3389/fgstr.2023.1245993